CLINICAL TRIAL: NCT04675619
Title: Evaluation of the Efficacy of Pirfenidone in Progressive Chronic Hypersensitivity Pneumonitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Eman Shebl, Assistant professor, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5889
Record Dates: First submitted 2020-12-11; First posted 2020-12-19 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: Hypersensitivity Pneumonitis
MeSH Terms: conditions — Alveolitis, Extrinsic Allergic | interventions — pirfenidone; Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral pirfenidone (Experimental): Pirfenidone will be administered orally in 267 mg capsules taken with food. The dose will be titrated over 2 weeks from one capsule three times a day during Week 1 to two capsules three times a day during Week 2 then maintenance dose (three capsules three times a day Week 3.
  Interventions: Drug: Oral pirfenidone
- Standard care (Experimental): Standard care
  Interventions: Drug: Standard care

INTERVENTIONS:
Drug: Oral pirfenidone — Treatment
  Arms: Oral pirfenidone
Drug: Standard care — Treatment
  Arms: Standard care

SUMMARY:
This study aims to evaluate the efficacy of pirfenidone in chronic hypersensitivity pneumonitis. This study included 40 adult patients (≥ 18 years) with a diagnosis of chronic progressive hypersensitivity pneumonitis. The included patients were divided into 2 groups 20 patients in each one.

Group 1: will receive pirfenidone in addition to the conventional treatment Group 2: will be maintained on conventional treatment. Forced vital capacity (FVC),6 minutes walking test(6MWT), oxygen tension in the arterial blood (PaO2), and St. George's Respiratory Questionnaire (SGRQ ) were measured before and after 6 months of a pirfenidone treatment trial.

Results

DETAILED DESCRIPTION:
Rationale The present data about the treatment of CHP are few and largely based on observational studies and expert opinion. It is suggested that pirfenidone may slow disease progression in cases of CHP as it has some anti-inflammatory in addition to antifibrotic effects.

Hypothesis Pirfenidone will slow disease progression in hypersensitivity pneumonitis patients

Research questions

1. Can pirfenidone slow disease progression in cases of CHP?
2. What about the safety of pirfenidone in cases of CHP?

This study aims to evaluate the efficacy of pirfenidone in chronic hypersensitivity pneumonitis.

Objectives

1. To compare the functional and radiological parameters between patients group who receive pirfenidone treatment and the patient group who receive conventional treatment: FVC, 6 minutes walking distance, the partial pressure of oxygen in arterial blood ( PaO2), Pulmonary artery systolic pressure, St.George's Respiratory Questionnaire(SGRQ Score) and Quantitative ILD score (QILD), by quantitative HRCT chest.
2. To compare the side effects between patients' group who receive pirfenidone treatment and the patient group who receive placebo treatment

Study design An interventional randomized controlled study

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old with a diagnosis of chronic progressive Hypersensitivity pneumonitis:
* >10% extent of fibrosis (eg, reticulation) on high-resolution CT (HRCT) scan
* Absolute decline in FVC% predicted >5% within the previous 6 months despite conventional treatment.

Exclusion Criteria:

* Pregnancy or breastfeeding period
* Patients with peptic ulcer, severe hepatic disease, severe kidney disease, severe cardiac disease, and patients with other chronic pulmonary diseases.
* Presence of active infection
* History of alcohol or drugs abuse
* Active smokers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Forced Vital Capacity (FVC) | Baseline to 6 months
  Forced vital capacity (FVC) is the volume of air that can forcibly be blown out after full inspiration,. FVC is the most basic maneuver in spirometry tests.
6 minutes walking distance | Baseline to 6 months
  The 6-min walk test (6MWT) has gained importance in the assessment of functional exercise capacity in patients with chronic respiratory disease.

CONTACTS AND LOCATIONS:
Locations (1):
- Eman Shebl, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cottin V, Hirani NA, Hotchkin DL, Nambiar AM, Ogura T, Otaola M, Skowasch D, Park JS, Poonyagariyagorn HK, Wuyts W, Wells AU. Presentation, diagnosis and clinical course of the spectrum of progressive-fibrosing interstitial lung diseases. Eur Respir Rev. 2018 Dec 21;27(150):180076. doi: 10.1183/16000617.0076-2018. Print 2018 Dec 31. PMID 30578335
- [Background] Li T, Guo L, Chen Z, Gu L, Sun F, Tan X, Chen S, Wang X, Ye S. Pirfenidone in patients with rapidly progressive interstitial lung disease associated with clinically amyopathic dermatomyositis. Sci Rep. 2016 Sep 12;6:33226. doi: 10.1038/srep33226. PMID 27615411